CLINICAL TRIAL: NCT01673282
Title: A Non-interventional, Observational Study Evaluating Changes in Drug Load and Seizure Frequency Using Vimpat (Lacosamide) in Daily Clinical Practice in Combination Therapy With Sodium Channel Blocking Anti-epileptic Drugs (AEDs) or Non Sodium Channel Blocking AEDs
Brief Title: Study Evaluating Changes in Total Drug Load and Seizure Frequency Using Vimpat® (Lacosamide) in Combination Therapy
Acronym: VICTOS
Status: Completed | Type: Observational
Sponsor: UCB Pharma GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: SP1065
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-09

CONDITIONS: Focal Epilepsy With and Without Secondary Generalization
Keywords: Lacosamide; Vimpat; Focal Epilepsy; Drug Load; AED; SP1065
MeSH Terms: conditions — Epilepsies, Partial | interventions — Lacosamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vimpat + Na Channel Blocking AED: Patients prescribed adjunctive lacosamide (LCM) added to one or more baseline Anti-Epileptic Drugs (AEDs) to include at least 1 sodium channel blocking AED.
  Interventions: Drug: Lacosamide
- Vimpat + Non-Na Channel Blocking AED: Patients prescribed adjunctive lacosamide (LCM) added to one or more baseline Anti-Epileptic Drugs (AEDs), none of which is a sodium channel blocking AED.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Route of Administration: oral/subcutaneous Form and Dosage: Tablet (50 mg/100 mg/150 mg, 200 mg); Syrup (10 mg/ml); Solution for infusion (10 mg/ml).
  Other Names: Vimpat; LCM

SUMMARY:
This observational study aims to investigate how VIMPAT® is used as adjunctive therapy in clinical practice and will also evaluate the subsequent change in the drug load of patients after addition of VIMPAT® to their treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* The patient has not received Vimpat® more than 7 days prior to start of Non-Interventional Study (NIS)
* The patient must have a diagnosis of epilepsy with partial-onset seizures with or without secondary generalization
* Based on the physician's clinical judgment, it is in the patient's best interest to be prescribed adjunctive Vimpat® (ie, the decision to prescribe Vimpat® is made by the physician)
* Patient must be at least 18 years of age
* The patient must have had at least one seizure within the last 3 months prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with focal epilepsy with or without secondary generalization.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (42):
- Austria (3):
  - 60, Innsbruck
  - 61, Mauer bei Amstetten
  - 63, Ried
- Germany (39):
  - 18, Berlin
  - 34, Berlin
  - 43, Berlin
  - 66, Berlin
  - 23, Bonn
  - 28, Cologne
  - 40, Cologne
  - 25, Dortmund
  - 35, Düsseldorf
  - 48, Erbach im Odenwald
  - 59, Erlangen
  - 30, Essen
  - 47, Giessen
  - 29, Göttingen
  - 37, Göttingen
  - 05, Haag
  - 12, Halle
  - 19, Halle
  - 39, Heidenheim
  - 54, Ibbenbueren
  - 27, Jena
  - 04, Jülich
  - 13, Kehl-Kork
  - 36, Kiel
  - 38, Leipzig
  - 52, Magdeburg
  - 67, Mainz
  - 49, Mittweida
  - 01, München
  - 08, Oranienburg
  - 17, Osnabrück
  - 14, Radeberg
  - 15, Rüsselsheim am Main
  - 16, Senftenberg
  - 41, Stuttgart
  - 09, Troisdorf
  - 22, Tübingen
  - 20, Ulm
  - 07, Westerstede

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in Austria and Germany in July 2012 and concluded in July 2015.
Pre-assignment Details: The Participant Flow consists of subjects in the Safety Set (SS) which received at least 1 dose of VIMPAT. Of the 315 enrolled subjects 311 were included in the SS.
Period: Overall Study
Arm/Group | Vimpat + Na Channel Blocking AED | Vimpat + Non-Na Channel Blocking AED
Started | 153 | 158
Completed | 120 | 132
Not Completed | 33 | 26
Not completed — Adverse Drug Reaction - Vimpat | 9 | 5
Not completed — Lack of Efficacy | 9 | 2
Not completed — Lost to Follow-up | 11 | 10
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Other | 1 | 6

BASELINE CHARACTERISTICS:
Population: The analysis group for Baseline Characteristics is the Safety Set (SS). The Safety Set consists of all patients who received at least 1 dose of Lacosamide.
Arm/Group | Vimpat + Na Channel Blocking AED | Vimpat + Non-Na Channel Blocking AED | Total Title
Number analyzed (Participants) | 153 | 158 | 311
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 135 | 117 | 252
  >=65 years | 17 | 41 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (16.4) | 52.5 (16.0) | 48.3 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 66 | 145
  Male | 74 | 92 | 166

OUTCOME MEASURES:

1. Primary Outcome: The Percent Change in Ratio of Dose and Defined Daily Dose (DDD) for the Drug Load of Concomitant Anti-Epileptic Drugs (AEDs) From Baseline to the End of Observation Period (Day 0 to 6 Months)
Description: Drug load is defined as the sum of the ratios of the actual doses divided by the defined daily dose for all concomitant AEDs.
Time Frame: From Baseline (Day 0) to 6 months
Population: The analysis group for the outcome measure is the Full Analysis Set (FAS). The FAS included all patients who received at least 1 dose of Lacosamide and for whom at least 1 valid ratio of dose and DDD at Baseline and post-Baseline could be calculated.
Measure: Mean (Standard Deviation); unit: percent change of ratio in dose
Arm/Group | Vimpat + Na Channel Blocking AED | Vimpat + Non-Na Channel Blocking AED
Number analyzed (Participants) | 149 | 153
percent change of ratio in dose | -15.0 (64.8) | -4.4 (31.9)
Statistical Analysis 1: Comparison: Vimpat + Na Channel Blocking AED vs Vimpat + Non-Na Channel Blocking AED; Based on an ANCOVA model for absolute change in ratio of dose and DDD with group as a fixed effect and the ratio of dose and DDD at Baseline as a covariate; Test type: Superiority or Other; p = 0.0003, ANCOVA; Least Square Mean = -0.24, 95% CI 2-sided [-0.36 to -0.11], Standard Error of Mean 0.06

ADVERSE EVENTS:
Time Frame: During the entire study period (day 0 - month 6)
Description: All patients who received at least 1 dose of Lacosamide were included in the SS.
Arm/Group | Vimpat + Na Channel Blocking AED | Vimpat + Non-Na Channel Blocking AED
Serious Adverse Events (participants affected / at risk) | 1/153 | 6/158
Other Adverse Events (participants affected / at risk) | 22/153 | 9/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vimpat + Na Channel Blocking AED (N=153) | Vimpat + Non-Na Channel Blocking AED (N=158)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Adverse event (General disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vimpat + Na Channel Blocking AED (N=153) | Vimpat + Non-Na Channel Blocking AED (N=158)
Drug ineffective (General disorders) | 9 (9) | 2 (2) — Adverse event terminology as reported by the investigator.
Off label use (Injury, poisoning and procedural complications) | 15 (16) | 7 (7) — Adverse event terminology as reported by the investigator.
Overdose (Injury, poisoning and procedural complications) | 15 (16) | 7 (7) — Overdose was defined as any Vimpat dose that was higher than the maximum approved dose of 400 mg/day. Adverse event terminology as reported by the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days